CLINICAL TRIAL: NCT00005254
Title: Natural History of Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1136; R01HL042973 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2000-06

CONDITIONS: Atherosclerosis; Coronary Disease; Arterial Occlusive Diseases; Peripheral Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Atherosclerosis; Coronary Disease; Arterial Occlusive Diseases; Peripheral Vascular Diseases; Cardiovascular Diseases

SUMMARY:
The Veterans Administration Patient Study examined the progression of peripheral arterial disease (PAD) in patients with large vessel PAD or isolated small vessel PAD. The Community Follow-up Study following subjects with and without PAD from a previous cohort to determine subsequent coronary heart disease and cardiovascular disease morbidity and mortality.

DETAILED DESCRIPTION:
BACKGROUND:

Peripheral arterial disease is a common condition, particularly in the elderly, but is the least frequently studied and the least well understood of the major atherosclerotic diseases.

DESIGN NARRATIVE:

Veterans Administration Patient Study: The progression of PAD was followed in patients diagnosed at the San Diego VA Medical Center from July 1984 to June 1989. Four non-invasive tests used in the initial diagnosis were repeated after a five year interval. The tests included segmental blood pressure flow velocity by Doppler ultrasound, post-occlusive reactive hyperemia, and pulse reappearance time. Risk factors examined for related to PAD included cigarette smoking, alcohol consumption, lipids and lipoproteins, blood pressure, fasting plasma glucose, diabetes history, immunoglobulin E, and creatinine. The degree of concordance between PAD and carotid disease was evaluated using phonoangiography.

Community Follow-up Study: The study was conducted in a cohort first examined for PAD in 1978-1981 and followed for morbidity and mortality.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-04; Study Completion 1995-03 (Actual)

REFERENCES:
- [Background] Criqui MH, Langer RD, Fronek A, Feigelson HS, Klauber MR, McCann TJ, Browner D. Mortality over a period of 10 years in patients with peripheral arterial disease. N Engl J Med. 1992 Feb 6;326(6):381-6. doi: 10.1056/NEJM199202063260605. PMID 1729621
- [Background] Criqui MH, Langer RD, Fronek A, Feigelson HS. Coronary disease and stroke in patients with large-vessel peripheral arterial disease. Drugs. 1991;42 Suppl 5:16-21. doi: 10.2165/00003495-199100425-00005. PMID 1726213
- [Background] Feigelson HS, Criqui MH, Fronek A, Langer RD, Molgaard CA. Screening for peripheral arterial disease: the sensitivity, specificity, and predictive value of noninvasive tests in a defined population. Am J Epidemiol. 1994 Sep 15;140(6):526-34. doi: 10.1093/oxfordjournals.aje.a117279. PMID 8067346
- [Background] Long TH, Criqui MH, Vasilevskis EE, Denenberg JO, Klauber MR, Fronek A. The correlation between the severity of peripheral arterial disease and carotid occlusive disease. Vasc Med. 1999;4(3):135-42. doi: 10.1177/1358836X9900400303. PMID 10512592
- [Background] Bird CE, Criqui MH, Fronek A, Denenberg JO, Klauber MR, Langer RD. Quantitative and qualitative progression of peripheral arterial disease by non-invasive testing. Vasc Med. 1999;4(1):15-21. doi: 10.1177/1358836X9900400103. PMID 10355865
- [Background] Criqui MH, Denenberg JO, Bird CE, Fronek A, Klauber MR, Langer RD. The correlation between symptoms and non-invasive test results in patients referred for peripheral arterial disease testing. Vasc Med. 1996;1(1):65-71. doi: 10.1177/1358863X9600100112. PMID 9546918